CLINICAL TRIAL: NCT06656468
Title: Outcome of Patients Undergoing Leadless Pacemaker Implantaton
Acronym: OPUPI
Status: Enrolling by invitation | Type: Observational
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Principal Investigator, Pietro Palmisano, Principal Investigator, Azienda Ospedaliera Cardinale G. Panico
Other Study IDs: OPUPI registry
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Bradyarrhythmias
Keywords: Bradyarrhythmias; leadless pacemaker; complications
MeSH Terms: conditions — Bradycardia | interventions — Defibrillators

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Leadless pacemaker patients: Consecutive patients undergoing leadless pacemaker patients
  Interventions: Device: Pacemaker and defibrillator

INTERVENTIONS:
Device: Pacemaker and defibrillator — Leadless pacemaker implantation procedure performed accordng to usual clinical practice. The indication for pacemaker implantation will be based on current guidelines.

SUMMARY:
Observational study aimed to evaluate the rate and of complications related to lealdless pacemaker implantation.

DETAILED DESCRIPTION:
Observational, multicenter study enrolling consecutive patients undergoing leadless pacemaker implantation. Procedure details, intraprocedural complications, and n-hospital outcomes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients with indication for leadless pacemaker implantation according to current Guidelines on cardiac pacing.

Exclusion Criteria:

* inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for leadless pacemaker implantation for symptomatic bradyarrhythmias according to current Guidelines on cardiac pacing.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Acute complications | From date of implantation until the date of first documented complication, assessed up to 30 days.
  Acute complications related to leadless pacemaker implantation

SECONDARY OUTCOMES:
Long-term complications | From 31th day from implantation until the date of first documented complication, assessed up to 6 months.
  Complications related to leadless pacemaker implantation observed during long-term follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera "Card. G. Panico", Tricase, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palmisano P, Facchin D, Ziacchi M, Nigro G, Nicosia A, Bongiorni MG, Tomasi L, Rossi A, De Filippo P, Sgarito G, Verlato R, Di Silvestro M, Iacopino S. Rate and nature of complications with leadless transcatheter pacemakers compared with transvenous pacemakers: results from an Italian multicentre large population analysis. Europace. 2023 Feb 8;25(1):112-120. doi: 10.1093/europace/euac112. PMID 36036679